CLINICAL TRIAL: NCT00953095
Title: Optimizing Social and Communication Outcomes for Young Children With Autism
Brief Title: Social and Communication Outcomes for Young Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Collaborators: University of California, Los Angeles (Other); University of Washington (Other); University of Michigan (Other); Florida State University (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Connie Kasari, Ph.D., Professor of Psychological Studies in Education and Psychiatry, Health Resources and Services Administration (HRSA)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: G09-02-016-01; UA3MC11055 (Other Grant/Funding Number: Health Resources and Services Administration)
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; treatment; joint attention; communication; language
MeSH Terms: conditions — Autism Spectrum Disorder; Communication; Language

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Caregiver Mediated Model (CMM) (Experimental): focuses on joint attention/engagement intervention using an established evidence based treatment (Kasari et al., 2006). It involves meeting the parent and child in their home for one hour, twice a week for 12 weeks. In this intervention, the parent-child pair meet with the interventionist (as opposed to the group training in the CEM condition). Parents will be specifically taught techniques for altering the home environment and ways to enhance children's language, social, and play development. Parents will given guided practice (input and coaching from the interventionist) as they implement these techniques with their child.
  Interventions: Behavioral: Joint Attention Intervention
- Caregiver Education Model (CEM) (Experimental): focuses on teaching parents information about autism, behavior modification, and community services using a manualized approach (Brereton & Tonge, 2005). Parents will receive information on child development each week, and will be able to ask questions and discuss the information vis-à-vis their own child. This intervention is manualized (Brereton & Tonge 2005). In the CEM condition, parents meet in a group (without their children) in a community-based setting to receive the intervention. Intervention sessions occur once a week for 2 hours.
  Interventions: Behavioral: Joint Attention Intervention

INTERVENTIONS:
Behavioral: Joint Attention Intervention — Intervention in both conditions occurs once a week for 2 hours. Participants will be randomized to 1 of 2 interventions : (1) Caregiver Mediated Model (CMM):focuses on joint attention/engagement and involves individual meetings with the parents and children at their homes. Parents will be specifically taught techniques for altering the home environment and ways to enhance children's language, social, and play development. Parents will given guided practice (input/ coaching from the interventionist) as they implement these techniques with their child. (2) Caregiver Education Model (CEM): focuses on teaching parents information about autism, behavior modification, and community services. Parents will receive information on child development each week, and will be able to ask questions and discuss the information. Parents meet in a group (without their children) in a community-based setting to receive the intervention.

SUMMARY:
The goal of this project is to test an intervention program for caregivers and their young children with autism that is focused on improving social communication. This study specifically targets underserved populations, specifically children from low SES and racial/ethnic minority families. Participants will include 40 children (aged 24 months to 60 months) and their caregivers who will be randomized (as if by flipping a coin) to one of the two treatments: Parent education sessions for two hours a week for 12 weeks or parent-child intervention sessions with the child for one hour, twice a week for 12 weeks. Young children with autism have difficulty with engaging in joint attention with others (e.g. pointing, showing. Joint attention skills are important to later development of language. Therefore, targeting this problem in young children may result in better language outcomes for these children.

In order to examine the effects of the interventions, all participants will be complete cognitive, language, communication and play-based assessments prior to treatment, at the end of the first 12 weeks of the intervention, and post-treatment immediately following the intervention (approximately 2.5 to 3 hours each).

DETAILED DESCRIPTION:
Child/parent dyads will be randomized to one of two intervention conditions: (1) Parent-child model, also known as the Caregiver Education Model (CMM):focuses on joint attention/engagement intervention using an established evidence based treatment (Kasari et al., 2006). It involves individual interventionist meetings with the parents and their children in their homes for one hour, twice a week for 12 weeks. In this intervention, the parent-child pair meet with the interventionist (as opposed to the group training in the CEM condition). Parents will be specifically taught techniques for altering the home environment and ways to enhance children's language, social, and play development. Parents will given guided practice (input and coaching from the interventionist) as they implement these techniques with their child. (2)Parent-education intervention, also known as the Caregiver Education Model (CEM): focuses on teaching parents information about autism, behavior modification, and community services using a manualized approach (Brereton & Tonge, 2005). Parents will receive information on child development each week, and will be able to ask questions and discuss the information vis-à-vis their own child. This intervention is manualized (Brereton & Tonge 2005). In the CEM condition, parents meet in a group, without their children, in a community-based setting to receive the intervention. Intervention in both conditions occurs for 2 hours for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Children must be between 24 months and 60 months at entry into the study
* Children must have a clinical diagnosis of autism or PDD-NOS, and/or meet criteria on the ADOS for ASD or autism
* Children must have an age equivalent of 12 months or greater for non-verbal ability based on the Mullen Visual Reception and Fine Motor scales
* Caregiver and child must be available for all assessments
* Children must be able to walk independently
* Parents must be between the ages of 16 and 50 years old
* Family should be currently underserved (inability to obtain services for their child) and have limited family resources

Exclusion Criteria:

* Children must not have a seizure disorder
* Children must not have associated sensory (uncorrected hearing loss greater than 20 db or vision loss) or physical disorders that restrict mobility (e.g., cerebral palsy)
* Children must not have sustained a head injury
* Children's diagnosis of autism spectrum disorder must not be comorbid with other medical syndromes (e.g., Tuberose Sclerosis, Neurofibromatosis, Down syndrome, fragile X) or diseases
* Children must not be in foster care
* English must be the primary language spoken at home
* Parents must not have a psychiatric diagnosis or a diagnosis of mental retardation

Ages: 24 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2009-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Early Social Communication Scale | Before treatment, after treatment and 3 months after treatment

SECONDARY OUTCOMES:
Mullen Scales of Early Learning | Before treatment, after treatment, and 3 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Connie Kasari, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (5):
- United States (5):
  - University of California, Los Angles, Los Angeles, California
  - Florida State University, Tallahassee, Florida
  - Kennedy Krieger Institute, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - University of Washington, Seattle, Washington

REFERENCES:
- [Background] Rutter M. Diagnosis and definition of childhood autism. J Autism Child Schizophr. 1978 Jun;8(2):139-61. doi: 10.1007/BF01537863. No abstract available. PMID 670129
- [Background] Mahoney, G., Kaiser, A., Girolametto, L., MacDonald, J., Robinson, C., Safford, P., & Spiker, D. (1999). Parent education in early intervention: A call for a renewed focus. Topics in Early Childhood Special Education, 19(3), 131-140.
- [Background] Koegel RL, Bimbela A, Schreibman L. Collateral effects of parent training on family interactions. J Autism Dev Disord. 1996 Jun;26(3):347-59. doi: 10.1007/BF02172479. PMID 8792265
- [Background] Kasari C, Freeman S, Paparella T. Joint attention and symbolic play in young children with autism: a randomized controlled intervention study. J Child Psychol Psychiatry. 2006 Jun;47(6):611-20. doi: 10.1111/j.1469-7610.2005.01567.x. PMID 16712638
- [Background] Whalen C, Schreibman L. Joint attention training for children with autism using behavior modification procedures. J Child Psychol Psychiatry. 2003 Mar;44(3):456-68. doi: 10.1111/1469-7610.00135. PMID 12635974
- [Background] Adamson LB, Bakeman R, Deckner DF, Romski M. Joint engagement and the emergence of language in children with autism and Down syndrome. J Autism Dev Disord. 2009 Jan;39(1):84-96. doi: 10.1007/s10803-008-0601-7. Epub 2008 Jun 26. PMID 18581223
- [Background] Tomasello M, Farrar MJ. Joint attention and early language. Child Dev. 1986 Dec;57(6):1454-63. PMID 3802971
- [Derived] Swain D, Li Y, Brown HR, Petkova E, Lord C, Rogers SJ, Estes A, Kasari C, Kim SH. Implementing a Uniform Outcome Measurement Approach for Early Interventions of Autism Spectrum Disorders. J Am Acad Child Adolesc Psychiatry. 2025 Jun;64(6):699-709. doi: 10.1016/j.jaac.2024.06.004. Epub 2024 Jul 2. PMID 38964630